CLINICAL TRIAL: NCT05742178
Title: NYC Cancer Outreach Network in Neighborhoods for Equity and Community Translation Randomized Controlled Trial (NYC CONNECT)
Brief Title: NYC Cancer Outreach Network in Neighborhoods for Equity and Community Translation
Acronym: NYC CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-01516
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer Screening
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (PN) (Experimental): Participants randomized to the PN arm will receive community health worker (CHW)-administered PN for cancer screening + social service needs + culturally and linguistically tailored cancer education. All individuals will complete a survey at baseline, 3 months, and 6 months.
  Interventions: Behavioral: Patient Navigation (PN) - More Intensive; Behavioral: Educational Materials
- Less Intensive (LI) (Active Comparator): Participants randomized to LI arm will receive PN to social service needs + culturally and linguistically tailored cancer education materials. All individuals will complete a survey at baseline, 3 months, and 6 months. Once a participant randomized to the LI arm completes the 6-month survey, they will have the option to receive all navigational support provided by CHWs to individuals randomized to the PN arm.
  Interventions: Behavioral: Educational Materials; Behavioral: Patient Navigation (PN) - Less Intensive

INTERVENTIONS:
Behavioral: Patient Navigation (PN) - More Intensive — The PN intervention will be administered by trained, bilingual CHWs: they will screen participants for cancer screening status and social needs and provide navigational support to cancer screening and social services.
  Arms: Patient Navigation (PN)
Behavioral: Educational Materials — Both PN and LI participants will receive tailored educational materials around cancer screening and SDH resources as needed.
Behavioral: Patient Navigation (PN) - Less Intensive — The PN intervention will be administered by trained, bilingual CHWs: they will screen participants for social needs and provide navigational support to social services.
  Arms: Less Intensive (LI)

SUMMARY:
NYC CONNECT will carry out a randomized controlled trial (RCT) which will assess the relative effectiveness of two evidence-based strategies to increase cancer screening rates for breast, cervical, and colorectal cancer. The RCT will compare the effectiveness of using a combination of 1) culturally and linguistically tailored cancer education materials and 2) community health workers (CHWs) to provide navigation services for cancer screening (the "patient navigation" [PN] arm) versus providing culturally and linguistically tailored cancer education only (the "less intensive" [LI] arm). The study population will include individuals who are due for breast, cervical, or colorectal cancer screening. All individuals recruited to the study will be provided navigation for unmet social determinants of health (SDH) needs.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 21 and 75 years;
* Men between the ages of 45 and 75 years;
* Women (40-74 years) who have not had a mammogram in the past 12 months, a Pap smear in the last 3 years (21-64 years old) or HPV test in the last 5 years (30-64 years old), or women 45-75 years old who are not up-to-date on colorectal cancer screening (Fecal occult blood test (FOBT)/Fecal immunochemical test (FIT) past year, computerized tomography (CT) colonography or sigmoidoscopy past 5 years, or colonoscopy past 10 years);
* Men not up-to-date on colorectal cancer screening (FOBT/FIT past year, computerized tomography (CT) colonography or sigmoidoscopy past 5 years, or colonoscopy past 10 years);
* Must speak either English, Spanish, Haitian-Creole, French, or Chinese (Mandarin and Cantonese);
* Lives in East Flatbush (zip codes: 11236, 11203, 11212, 11226); Sunset Park (zip codes: 11215, 11220, 11232); Highbridge (zip code 10452, 10455, 10451); or Morrisania (zip codes: 10456, 10459)

Exclusion Criteria:

* Previous or current diagnosis of any cancer;
* Pregnancy (breast and cervical cancer only);
* Current participation in an existing cancer navigation program;
* Currently in hospice care;
* At least 66 years of age with advanced illness or frailty or who live in long-term institution for more than 90 days;
* Bilateral mastectomy or right and left unilateral mastectomy (breast cancer only);
* Hysterectomy with no residual cervix (cervical cancer only);
* Total colectomy (colorectal cancer only).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Receive at Least 1 Cancer Screening at 6 Months After Study Enrollment | Up to Month 6
  Cancer screening defined as a breast, cervical, or colorectal cancer screening.

CONTACTS AND LOCATIONS:
Overall Officials: Chau Trinh, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Madison.LeCroy@nyulangone.org. Data will also be available for 5 years at a data repository, appropriately selected with the guidance of Nicole Contaxis, NYULH Data Catalog Coordinator. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Madison.LeCroy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. In addition, data will be available for 5 years at a data repository, appropriately selected with the guidance of Nicole Contaxis, NYULH Data Catalog Coordinator.
URL: https://datacatalog.med.nyu.edu/